CLINICAL TRIAL: NCT03475537
Title: The Usage of tDCS in Patients With Disorders of Consciousness
Brief Title: tDCS in Patients With Disorders of Consciousness
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: short of euqitments
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: test
Record Dates: First submitted 2018-03-18; First posted 2018-03-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2018-03

CONDITIONS: Consciousness Disorder; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Consciousness Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the treatment of transcranial direct current stimulation (Experimental): Direct current was applied by a battery-driven constant current stimulator using saline-soaked surface sponge electrodes (7×5 cm) with the anode positioned over the left dorsolateral prefrontal cortex (F3 according to the 10-20 international system for EEG placement) and the cathode placed over the right supraorbital region. During real tDCS, the current was increased to 2 mA from the onset of stimulation and applied for 20 minutes.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — the treatment of transcranial direct current stimulation

SUMMARY:
test

DETAILED DESCRIPTION:
Neurostimulation techniques such as deep brain stimulation (DBS) and spinal cord stimulation (SCS) have been used to treat DOC. Although these techniques have been shown to increase patient response, there are still some limitations. For example, DBS requires craniotomy and may increase the risk of intracranial hemorrhage and infection. In addition, the complexity and cost of these technologies also limit their potential applications.

ELIGIBILITY:
Inclusion Criteria:

Patients with DOC: VS and MCS (the cause of unification is: traumatic brain injury, the course of more than 1 month, not more than 1 year ; age 18-65; Past history without a mental disorder; No previous alcohol or substance abuse; No epilepsy or frequent spontaneous movement; No benzodiazepines; No moderate or severe hydrocephalus, All patients were right handed.

Exclusion Criteria:

Exclusion of organic heart disease, such as sinus bradycardia, arrhythmia; exclusion of patients with intracranial metal devices, pacemakers or any other device.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-15 (Estimated); Primary Completion 2019-07-15 (Estimated); Study Completion 2020-01-15 (Estimated)

PRIMARY OUTCOMES:
improvement of CRS-R | 7 days
  test

CONTACTS AND LOCATIONS:
Overall Officials: Benyan Luo, Principal Investigator — Department of Neurology and Brain Medical Centre The First Affiliated Hospital, School of Medicine, Zhejiang University 79 Qingchun Road, Hangzhou
Locations (1):
- The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided